CLINICAL TRIAL: NCT06038461
Title: An Open, Single-center Clinical Study of Surufatinib Combined With Temozolomide and S-1 in the First-line Treatment of Advanced Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yihebali Chi, MD, Professor, Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-NEN106
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Tumors
Keywords: Surufatinib; Temozolomide and S-1; First-line treatment
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Temozolomide; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Surufatinib Combined With Temozolomide and S-1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib Combined With Temozolomide and S-1 (Experimental): Patients will receive surufatinib combined with temozolomide and S-1 once every three weeks as the second-line treatment until disease progression or intolerable toxicity or patients withdrawal of consent.
  Phase I: DLTs of surufatinib combined with temozolomide and S-1 will be evaluated based on NCI CTCAE v 5.0 in the first cycle.
  Interventions: Drug: Surufatinib Combined With Temozolomide and S-1

INTERVENTIONS:
Drug: Surufatinib Combined With Temozolomide and S-1 — Phase I:
  Surufatinib: 250mg, QD, PO, Q3W; Temozolomide: 200-300mg, d10-d14, QD, PO, Q3W; S-1: 40-60mg, d1-d14, BID, PO, Q3W.
  Phase II:
  Surufatinib, Temozolomide and S-1：RP2D

SUMMARY:
This is a prospective, open, single-center study evaluating the efficacy and safety of surufatinib Combined With Temozolomide and S-1 as the first-line treatment of advanced neuroendocrine tumors

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75years (inclusive);
* Histopathologically confirmed diagnosis of advanced MGMT0/1+ (G1, G2 or G3) neuroendocrine tumor (locally advanced, unresectable or distant metastasis);
* Previously untreated with systemic therapy;
* Have at least one measurable lesion according to RECIST v1.1;
* ECOG performance status: 0-2(determined by investigator);
* Expected survival time > 3 months;
* Adequate hepatic, renal, heart, and hematologic functions;
* Urine protein < ++ . If Urine protein ≥ ++ ,the amount of urine protein in 24 hours ≤1.0g;
* Before the first dose, serum HCG examination of potential childbearing-women must be negative; Men/Women of childbearing potential must agree to use a highly effective contraceptive method (such as double barrier contraceptive method, condom, oral or injectable contraceptives and intrauterine device) throughout treatment and for at least 90 days after study completion.

Exclusion Criteria:

* Neuroendocrine cancer, adenocarcinoid, goblet cell carcinoid,
* Functional NETs which need to control symptoms by long-acting somatostatin analogues;
* Received a major surgery which requires at least 3 weeks after recovery time, to undergo surgery on treatment of this research within 4 weeks prior to treatment;
* Have uncontrolled hypertension, defined as systolic blood pressure >140 mmHg or diastolic blood pressure >90 mm Hg, while under anti-hypertension treatment;
* Patients with active ulcer, intestinal perforation and intestinal obstruction;
* With active bleeding or bleeding tendency;
* Severe history of cardiovascular and cerebrovascular diseases;
* Other malignancies diagnosed within the previous 5 years, except basal cell carcinoma or cervical carcinoma in situ after radical resection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | approximately 1 years
  the proportion of patients with complete response or partial response, using RESIST v1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | approximately 1 years
  time from first-dose to the first documented disease progression or death
Disease Control Rate (DCR) | approximately 1 years
  the proportion of patients with complete response, partial response or stable disease, using RESIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China